CLINICAL TRIAL: NCT01530360
Title: Safeguarding the Brains of Our Smallest Children - a Pilot Study
Brief Title: Cerebral Oxygenation to Guide Medical Interventions in Extremely Preterm Infants
Acronym: SafeBoosC-p
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Gorm Greisen (Other)
Collaborators: Elsass Foundation (Other); Copenhagen Trial Unit, Center for Clinical Intervention Research (Other); Medical University of Graz (Other); Hospices Civils de Lyon (Other); KU Leuven (Other); University College Cork (Other); University of Zurich (Other); University of Milan (Other); Universitair Medisch Centrum Utrecht (Unknown); University of Witten/Herdecke (Other); Uppsala University (Other); Cambridge University Hospitals NHS Foundation Trust (Other); Hospital Universitario La Paz (Other)
Responsible Party: Sponsor-Investigator, Gorm Greisen, professor,head of department, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: SBP010911
Record Dates: First submitted 2012-02-07; First posted 2012-02-09 (Estimated); Last update posted 2012-12-10 (Estimated); Status verified 2012-12

CONDITIONS: Premature Infants; Near-infrared Spectroscopy; Oximetry
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- cerebral oximetry + treatment guideline (Experimental): Cerebral oximetry applied as soon as possible after birth and continued until 72 hours of life Clinical staff administer the routine medical management according to local practice as well as respond to out-of-range values with the help of the treatment guideline
  Interventions: Device: cerebral oximeter

INTERVENTIONS:
Device: cerebral oximeter — INVOS 5100c + SAFB-SM SOMASENSOR NONIN EQUANOX 7600 + sensor model 8000CA

SUMMARY:
Regional tissue oxygenation (rStO2) can be monitored by near-infrared spectroscopy. The investigators planned a SafeBoosC phase II trial to test if a reduction of the burden of hyper- and hypoxia can be accomplished during the first three days of life in infants born before 28 completed weeks of gestation. The investigators developed a treatment guideline and a randomised trial design to evaluate if cerebral rStO2 spent out of range in %hours can be reduced by 50%. The present trial is a non-randomised pilot study of the intervention in 10 infants.

ELIGIBILITY:
Inclusion Criteria:

* gestational age at birth less than 28 completed weeks
* cerebral oximeter in place at 3 hours after birth

Exclusion Criteria:

* decision not to provide full life support

Max Age: 3 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 2011-09; Primary Completion 2011-12 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
change of medical management elicited by cerebral oxygenation out of range | 0-72 hours of life
  Recording of the type of change of management as defined by the treatment guideline

SECONDARY OUTCOMES:
Adverse device effects | 0-72 hours
  Expected and unexpected
burden of hypo-and hyperoxia | 0-72 hours
  measured as %hours out of the target range (55-85%)

CONTACTS AND LOCATIONS:
Overall Officials: Gorm Greisen, MD,DMSci, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Department of Neonatology, Rigshospitalet, Copenhagen, Denmark

REFERENCES:
- [Background] Greisen G, Leung T, Wolf M. Has the time come to use near-infrared spectroscopy as a routine clinical tool in preterm infants undergoing intensive care? Philos Trans A Math Phys Eng Sci. 2011 Nov 28;369(1955):4440-51. doi: 10.1098/rsta.2011.0261. PMID 22006900
- [Derived] Hyttel-Sorensen S, Austin T, van Bel F, Benders M, Claris O, Dempsey EM, Fumagalli M, Gluud C, Hagmann C, Hellstrom-Westas L, Lemmers P, Naulaers G, van Oeveren W, Pellicer A, Pichler G, Roll C, Stoy LS, Wolf M, Greisen G. Clinical use of cerebral oximetry in extremely preterm infants is feasible. Dan Med J. 2013 Jan;60(1):A4533. PMID 23340184